CLINICAL TRIAL: NCT06534827
Title: Investigating an Innovative Mentoring Model for Improving Effectiveness and Equity of Community-Based Support for Youth From Low-Resource Families With Mental Health Challenges
Brief Title: Study of Mental Health and Relationships
Acronym: SMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Herrera Consulting Group, LLC (Unknown)
Responsible Party: Principal Investigator, David DuBois, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 107309
Record Dates: First submitted 2024-03-01; First posted 2024-08-02 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Mental Health
Keywords: mentoring; mental health; youth; low-income; mental health interventions
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Services as Usual (No Intervention): Outpatient mental health services as usual
- GLM + Services as Usual (Experimental): The Great Life Mentoring program (GLM) provides volunteer-based mentoring for school-age youth from low-resource families who are receiving outpatient mental health care. Each youth is paired with a mentor with whom they spend time in the community on a weekly basis for at least one year. Mentors are required to complete a 20-hour intensive training prior to being paired with a youth. Mentors also receive monthly in-person supervision from GLM staff for the first year of their meetings, which continues on an as-needed basis thereafter. Training and supervision are geared toward the unique opportunities and challenges that can occur when mentoring a youth with mental health needs. The goal is for the mentor to become an integral part of the child's mental health treatment, but the mentoring relationship is also sustained after treatment ends.
  Interventions: Behavioral: Great Life Mentoring

INTERVENTIONS:
Behavioral: Great Life Mentoring — The Great Life Mentoring program (GLM) provides volunteer-based mentoring for school-age youth from low-resource families who are receiving outpatient mental health care. Each youth is paired with a mentor with whom they spend time in the community on a weekly basis for at least one year. Mentors are required to complete a 20-hour intensive training prior to being paired with a youth. Mentors also receive monthly in-person supervision from GLM staff for the first year of their meetings, which continues on an as-needed basis thereafter. Training and supervision are geared toward the unique opportunities and challenges that can occur when mentoring a youth with mental health needs. The goal is for the mentor to become an integral part of the child's mental health treatment, but the mentoring relationship is also sustained after treatment ends.
  Arms: GLM + Services as Usual

SUMMARY:
The goal of this clinical trial is to test effects of the Great Life Mentoring (GLM) program on the mental health and adaptive functioning on school-age youth (ages 9-16) from low-income families who are receiving outpatient mental health services. The main questions it aims to answer are:

• Does participation in the GLM program improve mental health and related outcomes among school-age youth (9- to 16-years-old) from low-income families as an adjunct to outpatient mental health services? 180 youth will be enrolled in the study and assigned randomly to either continue mental health services as usual (SAU) or to continue mental health services while also participating in GLM (SAU+GLM). Participating youth, and their parent/guardians and therapists, will be surveyed annually. Mental health services records also will be obtained with appropriate permissions. . Researchers will compare the SAU and SAU+GLM groups to see if participation in GLM has an effect on the mental health and related outcomes of study youth.

ELIGIBILITY:
Inclusion Criteria:

* Youth is between 9- and 16-years-old
* Youth meets eligibility criteria for the Great Life Mentoring program, which include receiving publically-subsidized outpatient mental health care

Exclusion Criteria:

* Parental primary language other than English
* Youth difficulties in cognitive functioning that would preclude ability to complete study assessments

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Mental Health | Annually throughout duration of study participation, average of 2 years
  Average of standardized (z-scored) scores on following study outcome measures:
  Depressive Symptoms (inverted), Anxiety Symptoms (inverted), Loneliness (inverted), Internalizing Symptoms (inverted), Externalizing Symptoms (inverted), Suicidal Ideation, Happiness, Life Satisfaction, Self-Esteem, and Hope
Depressive Symptoms | Annually throughout duration of study participation, average of 2 years
  Total raw score on the PROMIS (Patient-Reported Outcomes Measurement Information System) Pediatric Short-Form v2.0 Depressive Symptoms (8 items; youth self-report)
Anxiety Symptoms | Annually throughout duration of study participation, average of 2 years
  Total raw score on the PROMIS Pediatric Short-Form v2.0 Anxiety (8 items; youth self-report)
Loneliness | Annually throughout duration of study participation, average of 2 years
  Total raw score on NIH (National Institutes of Health) Toolbox Loneliness Fixed Form Ages 8-17 v2.0 (7 items; youth self-report)
Internalizing Symptoms | Annually throughout duration of study participation, average of 2 years
  Average of standardized (z-scored) Total scores on the Internalizing scale of the youth self-report and parent-report versions of the Symptoms and Functioning Severity Scale (SFSS) - Peabody Treatment Progress Inventory
Externalizing Symptoms | Annually throughout duration of study participation, average of 2 years
  Average of standardized (z-scored) Total scores on the Externalizing scale of the youth self-report and parent report versions of the Symptoms and Functioning Severity Scale (SFSS) - Peabody Treatment Progress Inventory
Life Satisfaction | Annually throughout duration of study participation,average of 2 years
  Total score on Brief Multidimensional Students' Life Satisfaction Scale (6 items; youth self-report)
Happiness | Annually throughout duration of study participation, average of 2 years
  Total raw score on PROMIS Pediatric Short Form v1.0 - Positive Affect 4a (4 items; youth self-report)
Suicidal Ideation | Annually throughout duration of study participation, average of 2 years
  Affirmative response on Youth Risk Behavior Surveillance item asking about suicidal ideation, tailored to refer to the past year (youth self-report)
Self-esteem | Annually throughout duration of study participation, average of 2 years
  Total score on Global Self-Esteem scale of the short-form of the Self-Esteem Questionnaire (4 items; youth self-report)
Hope | Annually throughout duration of study participation, average of 2 years
  Total score on abbreviated "Toolbox" version of the Hopeful Future Expectations Scale (7 items; youth self-report)

SECONDARY OUTCOMES:
Engagement in Mental Health Services | End of study participation, average of 2 years
  Percentage of scheduled mental health services sessions attended as indicated by mental health service records
Therapist-Youth Alliance | Annually throughout duration of study participation while youth is receiving mental health services, average of 1 year
  Average of standardized (z-scored) scores on therapist and youth report versions of the Therapist Alliance Scale for Children-Revised
Resilience | Annually throughout duration of study participation, average of 2 years
  Total score on The Resilience Scale (RS-14) (14 items; youth self-report)
Adaptive Coping with Stress | Annually throughout duration of study participation, average of 2 years
  Rating on single-item youth-report measure adapted from Coping Efficacy Scale (Sandler et al., 2000)
Emotion Regulation | Annually throughout duration of study participation, average of 2 years
  Total score on measure adapted from Prior et al. (2000) (4 items; youth self-report)
Empathy | Annually throughout duration of study participation, average of 2 years
  Total score on measure used in evaluation by Boys and Girls Clubs of America (4 items; youth self-report)
Spark (hobby/interest) | Annually throughout duration of study participation, average of 2 years
  Response on single item youth-report measure adapted from Search Institute Thriving Orientation Survey
Self-advocacy | Annually throughout duration of study participation,average of 2 years
  Total score on Self-advocacy Scale from Mentoring Enhancement Demonstration Project (4 items; youth self-report)
Goal-setting | Annually throughout duration of study participation, average of 2 years
  Average of standardized (z-scored) Total scores on Goal-setting scale from Kuperminc et al. (2011) (4 items; youth self-report) and the Goal Orientation Scale (Child Trends, 2022) (7 items, parent report)
Problem-solving | Annually throughout duration of study participation, average of 2 years
  Total score on Scale from Raising Healthy Children Survey (4 items; youth self-report)
Communication Skills | Annually throughout duration of study participation, average of 2 years
  Total score on measure used in evaluation by Boys and Girls Clubs of America (4 items; youth self-report)
Grit - Perseverance | Annually throughout duration of study participation, average of 2 years
  Total score on Perseverance subscale of the Short Grit Scale for Children (4 items, youth self-report0
Peer Social Skills | Annually throughout duration of study participation, average of 2 years
  Total score on Social Competence Sale of the Youth Outcome Measures Toolbox (7 items, youth self-report)
Social Support from Family | Annually throughout duration of study participation, average of 2 years
  Total score on Family subscale of the Multidimensional Scale of Perceived Social Support (4 items, youth self-report)
Social Support from Non-Parental Adults | Annually throughout duration of study participation, average of 2 years
  Total score on Special Persons subscale of the Multidimensional Scale of Perceived Social Support with items modified to refer to "special adult outside of my family" rather than "special person" (4 items, youth self-report)
Social Support from Peers | Annually throughout duration of study participation, average of 2 years
  Response on a single item developed for this study asking about whether the youth has a good friend around the same age (youth self-report)
Very Important Nonfamilial Adult | Annually throughout duration of study participation, average of 2 years
  Response on single item from DuBois et al. (2022) asking whether the youth has a very important adult in their life and, if so, in what category(ies), with endorsement of a category other than parent/primary caregiver or relative scored as 1 and other responses scored as 0. Other responses will be coded for applicability to the predetermined categories by persons blind to study arm.
Academic Success | Annually throughout duration of study participation, average of 2 years
  Response on single item from DuBois et al. (2022) asking about grades in school (youth self-report)
School Connectedness | Annually throughout duration of study participation, average of 2 years
  Total score on School subscale of Hemingway Measure of Adolescent Connectedness (6 items, youth self-report)
Career Exploration | Annually throughout duration of study participation, average of 2 years
  Total score on Future Planning: Talk to an Adult scale from the SAYO (Survey of Academic and Youth Outcomes)-Y (4 items, youth self-report)
Perceptions of Treatment Progress | Annually throughout duration of study participation, average of 2 years
  Average of standardized (z-scores) Total scores on youth- and parent-report versions Treatment Outcome Expectations Scale from the Peabody Treatment Progress Battery, with items modified to also refer to progress currently observed, not only expected (8 items)
Perceptions of Counseling Impact | Annually throughout duration of study participation while youth is receiving mental health services, average of 1 year
  Total score on adapted version of the Youth Counseling Impact Scale from the Peabody Treatment Progress Battery, with items modified to refer to last 2 weeks rather than a single session, 2 items added, and 3 items dropped (5 items)
Parent Stress | Annually throughout duration of study participation, average of 2 years
  Total score on measure from Pearlin & Schooler (1978) (11 items, parent-report)
Family Functioning | Annually throughout duration of study participation, average of 2 years
  Total score on General Functioning subscale of the Family Assessment Device (Epstein et al., 1983) (12 items, parent-report)
Positive Parenting | Annually throughout duration of study participation, average of 2 years
  Total score on Positive Parenting subscale of the Alabama Parenting Questionnaire (6 items, parent-report)
Parental Involvement | Annually throughout duration of study participation, average of 2 years
  Total score on Involvement subscale of the Alabama Parenting Questionnaire (10 items, parent-report)
Parental Poor Supervision | Annually throughout duration of study participation, average of 2 years
  Total score on Poor Monitoring/Supervision subscale of the Alabama Parenting Questionnaire (10 items, parent-report)
Self-Control | Annually throughout duration of study participation, average of 2 years
  Total score on Child Self-Control scale (Grasmick et al., 1993) (8 items, parent-report)
Social-emotional Learning Skills | Annually throughout duration of study participation, average of 2 years
  Total score on measure of student social and emotional competencies (Collaborative for Academic, Social, and Emotional Learning & the American Institutes for Research, 2013) (20 items, parent report)
Parent Depressive Symptoms | Annually throughout duration of study participation, average of 2 years
  Total raw score on PROMIS Short Form v1.0 - Depression 4a (4 items, parent self-report)
Parent Positive Affect | Annually throughout duration of study participation, average of 2 years
  Total raw score on PROMIS Pediatric Short Form v1.0 - Positive Affect 4a (4 items; parent self-report)
Parent-Child Alliance | Annually throughout duration of study participation, average of 2 years
  Total score on measure from the National Survey of Children's Health (5 items; parent report)
Successful Completion of Treatment | Point in time when youth's mental health treatment ends, average of 1 year
  Planned ending of treatment as determined by mental health records coded as 1 and unplanned, client-initiated ending, and endings for other reasons coded as 0.

CONTACTS AND LOCATIONS:
Overall Officials: David DuBois, PhD, Principal Investigator — University of Illinois Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of Great Life Mentoring program — http://greatlifementoring.com/